CLINICAL TRIAL: NCT04496700
Title: Transfusion of Whole Blood to Military Forces in a Combat Situation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010/1559
Record Dates: First submitted 2013-07-07; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2013-07

CONDITIONS: Autologous Blood Transfusion; Physical Performance; Donor Safety
Keywords: Autologous Blood Transfusion; Whole Blood Storage Conditions; Physical Performance; Donor Safety; Combat Field
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Intervention Model Description: The participants will take part in one of three tasks, and will be tested in their respective task twice: both before and after blood donation (the intervention).
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 - Shooting test (Experimental): All participants in this group were tested for shooting abilities before and after blood donation. No variation within the group.
  Interventions: Procedure: Whole blood donation and transfusion
- Group 2 - VO2max (Experimental): All participants in this group were tested for physical abilities before and after blood donation. Method: Bruce protocol.
  No variation of protocol within the group.
  Interventions: Procedure: Whole blood donation and transfusion
- Group 3 - Feasability (Experimental): All participants in this group were tested for feasability before and after blood donation. Method: Hiking uphill with 20 kg backpack.
  No variation of method within the group.
  Interventions: Procedure: Whole blood donation and transfusion

INTERVENTIONS:
Procedure: Whole blood donation and transfusion — The effect of whole blood donation on physical performance:
  Donation of 450 ml whole blood - one time only.

SUMMARY:
During military action there might be situations where civil requirements for blood transfusion are not obtainable. Numerous warfare experiences suggest that administration of whole blood to a patient with uncontrollable bleeding/bleeding shock will improve survival in case of delayed evacuation.

Among Norwegian troops this gives one of two choices:

1. A soldier donates blood to a wounded fellow soldier
2. Personnel in safe distance donates blood and it is transported to the frontline.

Alternative b might implicate frequent donations and unused blood must be auto-re-transfused.

This study will investigate:

1. Can 'buddy transfusion' in the field be justified also in medical aspects?
2. Can repeated donations and auto-transfusions of transported whole blood into personnel(X) be justified also in medical aspects?

(X) Blood typed and screened for HIV, HBV, HCV, Syphilis before assignment

DETAILED DESCRIPTION:
MATERIALS AND METHODS

The study was approved by the research ethics committee of the Regional West Health Trust, Norway. Twenty-five nonsmoking male soldiers, median age 29 years, from a Navy special forces unit consented to participate. Mean body mass index was 24.7 kg/m2 (range, 22.6-28.3 kg/m2).

This is a pilot study and we were not able to find data in the literature providing information for power calculations regarding the testing we included in the study. The participants were divided in three different groups for testing. The grouping was based on availability at the given time points, and there was no selection to any specific group: Group 1-Bruce protocol treadmill stress test, push-ups, and pull-ups (n = 7); Group 2-50-round pistol shooting test (n = 12); and Group 3-uphill hiking exercise carrying a 20-kg backpack (n = 6). Each group was tested twice, before and immediately after donation of 450 mL of blood.

The soldiers were allowed to rehydrate during the donation procedure and theywere all offered a 0.5-L water bottle. The exact volume each participant consumed was not recorded. All 25 soldiers participated in a 60-minute training program aimed at testing whether it is possible to teach nonmedic soldiers buddy transfusion during a short period.

Multistage treadmill stress test, push-ups, and pull-ups

VO2 max was estimated in seven soldiers. Bruce protocol was followed, using a multistaged treadmill test. Each stage lasted for 3 minutes, and in total seven stages were included in the procedure. For each stage, belt velocity and slope were increased (see Table 1). The soldiers ran until exhaustion (unable to continue running). Heart rate and lactate were measured at the end of each stage and at exhaustion when total time on belt (T) was noted. Lactate was measured in a blood sample from the ear lobule and a portable lactate analyzer (Lactate Scout, EKF Diagnostics, Barleben, Germany) was used. From the total run time used, VO2 max was estimated as follows:14 VO2 max = 14.8-(1.379 ¥ T) + (0.451 ¥ T2) - (0.012 ¥ T3). The pushups were performed as "full push-up" in the prone position, with the back and legs straight and off the floor. The hands were placed below each shoulder, with arms fully extended. From this start position, the body was lowered by using the arms until the chest touched the floor, and then back to the start position. Standard pull-ups were performed as a dead-hang pull-up, with an overhand grip. Then the body was pulled up until the chin cleared the bar, and finished by lowering the body until arms and shoulders were fully extended A baseline test (predonation test) was performed 4 days prior to donation, and the postdonation test immediately after donating blood. The soldiers performed the procedures until they were unable to continue. The test endpoint was differences in estimated VO2 max, maximum heart rate (HRmax), lactate, and number of push-ups and pull-ups.

Fifty-round pistol shooting test

Twelve soldiers performed a standard Navy special operational forces protocol rapid shooting test, using their personalweapon (9 mm).The protocol has five separate tests, each with 10 rounds (6 mnondominant hand, 10 mdominant hand, 10 m 2 + 1, 18 m precision, 25 m precision). The predonation test was performed 2 days before donation, and the postdonation test immediately after donating blood. The weather and light conditions were similar on the test days. The study outcome in this exercise was differences in total hits.

Uphill hiking exercise

Six soldiers were tested on an uphill exercise carrying a 20-kg backpack. The track had a 28% slope and 450-m altitude difference; the soldiers were instructed to walk as a group, and no individual time measurements could therefore be recorded. The soldiers walked up and down again as quickly as they were able to (no running) before they donated 1 unit of blood. They thenwere offered water (ad libitum) to rehydrate without any further break before they repeated the exercise, again walking as quickly as the group managed. The endpoint was the difference in time used by the team on the uphill part of the track. The soldiers also filled in a questionnaire to report possible side effects related to the donation and the postdonation performance.

ELIGIBILITY:
Inclusion Criteria:

* Military personel deployable to combat situations

Exclusion Criteria:

* General health issues

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of hits | Pre- and postdonation
  The effect of whole blood donation on Combat Readiness Skills is evaluated by various tasks, among them a 50-round pistol shooting test (Standard Navy SOF protocol). The shooting test was performed before and immediately after donation of 450 ml whole blood.
  This outcome measure depicts number of hits in total, pre- and postdonation, respectively.

SECONDARY OUTCOMES:
Maximum heart rate (n/min) | Pre- and postdonation
  The effect of whole blood donation on Combat Readiness Skills is evaluated by various tasks, among them a so-called Bruce protocol. This protocol was performed before and immediately after donation of 450 ml whole blood.
  This outcome measure depicts maximum heart rate (n per minute), pre- and postdonation, respectively.
Minutes spent walking up and down the mountain Ulriken | Pre- and postdonation
  The effect of whole blood donation on Combat Readiness Skills is evaluated by various tasks, among them hiking up and down a mountain with a 28 % slope, 450 meters altitude difference and a 20 kg backpack.
  The endurance test was performed before and immediately after donation of 450 ml whole blood.
  This outcome measure depicts time in minutes, spent walking up and down the moutain, pre- and postdonation, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Geir Strandenes, OF3, Principal Investigator — Haukeland UH
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Norwegian Naval Base Haakonsvern, Bergen